CLINICAL TRIAL: NCT03079622
Title: Manual Versus Electric Vacuum Aspiration for Pregnancy Termination Between 10-14 Weeks: A Randomized Trial
Brief Title: Manual Versus Electric Vacuum Aspiration for Pregnancy Termination Between 10-14 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2015-11-18; First posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Abortion in First Trimester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electric vacuum aspiration (Active Comparator): Electric vacuum aspiration will be performed with Synevac® Vacuum Curettage System 10 (Richmond, CA, USA) with a rigid cannula.
  Interventions: Procedure: Electric Vacuum Aspiration
- Manual vacuum aspiration (Active Comparator): Manual vacuum aspiration will be performed using the 60-mL double valve aspirator, manufactured by Ipas (Chapel Hill, NC, USA) with a flexible cannula.
  Interventions: Procedure: Manual Vacuum Aspiration

INTERVENTIONS:
Procedure: Electric Vacuum Aspiration
  Other Names: Synevac® Vacuum Curettage System 10
  Arms: Electric vacuum aspiration
Procedure: Manual Vacuum Aspiration
  Other Names: Ipas 60-mL double valve aspirator
  Arms: Manual vacuum aspiration

SUMMARY:
The study titled, Manual Versus Electric Vacuum Aspiration for Pregnancy Termination Between 10-14 weeks: A Randomized Trial, is a randomized trial to compare procedure times for manual and electric vacuum aspiration for surgical abortion between 10 0/7 and 13 6/7 weeks gestation. Women presenting for surgical abortion between 10 0/7 and 13 6/7 weeks gestation will be randomized to either undergo manual vacuum aspiration (MVA) or electric vacuum aspiration (EVA). The investigators hypothesize that operative times will be increased when using manual vacuum aspiration, as compared to electric vacuum aspiration, for surgical abortion performed in the late first trimester (10 0/7 and-13 6/7 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Between 10 0/7 and 13 6/7 weeks of gestation
* Documented intra-uterine pregnancy
* Presenting for surgical induced abortion at RHS
* English-speaking
* Age 18 or older

Exclusion Criteria:

* Spontaneous abortion
* Failed medical abortion
* Multiple gestation
* Uterine anomalies
* Lower uterine segment or cervical myomas
* History of 3 or more prior cesarean deliveries
* BMI > 40
* Having the abortion procedure performed by a provider who does not perform MVA and EVA between 10 0/7 and 13 6/7 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Operative time | Perioperative
  Time from cannula insertion until completion of uterine evacuation

SECONDARY OUTCOMES:
Conversion from electric to manual vacuum aspiration (or vice versa) during the procedure | Perioperative
Provider acceptability | Perioperative
  1) Ease of procedure on a 5 point Likert scale, 2) Appropriateness of method used for procedure (binary response)
Patient acceptability | Perioperative and 2 weeks postoperatively
  1) Satisfaction with procedure on 4-point rating scale 2) Would choose same procedure again (binary response) 3) Would recommend procedure to a friend (binary response)

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn M Grentzer, MD, MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data, except de-identified data within our division.